CLINICAL TRIAL: NCT07333170
Title: Comparison of the Efficacy of Topical Luliconazole 2% Cream vs Topical Ketoconazole 1% Cream in the Treatment of Pityriasis Versicolor.
Acronym: P versicolor
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: PAEC General Hospital, Islamabad (Other)
Collaborators: PAEC general hospital (Other Government)
Responsible Party: Principal Investigator, Sana Rafique, Post graduate trainee, PAEC General Hospital, Islamabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAECIslamabad
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pityriasis Versicolor
Keywords: P versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — Ketoconazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. One group will receive topical luliconazole, while the other group will receive topical ketoconazole for the treatment of pityriasis versicolor. Clinical and mycological outcomes will be compared between the two groups.
Masking Description: This is an open-label study; no participants, care providers, investigators, or outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Luliconazole 1% cream (Experimental): Participants will receive topical luliconazole 1% cream applied once daily to affected areas for the treatment of pityriasis versicolor.
  Interventions: Drug: Luliconazole Cream 1%
- Topical ketoconazole 2% cream (Experimental): Participants will receive topical ketoconazole 2% cream applied twice daily to affected areas for the treatment of pityriasis versicolor.
  Interventions: Drug: Topical ketoconazole 2% cream

INTERVENTIONS:
Drug: Luliconazole Cream 1% — Ketoconazole is relatively hydrophilic with limited skin retention, whereas luliconazole is highly lipophilic, resulting in superior stratum corneum penetration, higher keratin binding, and prolonged antifungal activity.
  Arms: Topical Luliconazole 1% cream
Drug: Topical ketoconazole 2% cream — Ketoconazole is relatively hydrophilic with limited skin retention, whereas luliconazole is highly lipophilic, resulting in superior stratum corneum penetration, higher keratin binding, and prolonged antifungal activity.
  Arms: Topical ketoconazole 2% cream

SUMMARY:
Pityriasis versicolor is a common superficial fungal infection caused by Malassezia species, characterized by hypo- or hyper-pigmented scaly patches on the skin. Topical antifungal agents are the mainstay of treatment. Ketoconazole has been widely used; however, newer agents such as luliconazole may offer improved efficacy and shorter treatment duration. This randomized controlled study aims to compare the efficacy and safety of topical luliconazole versus topical ketoconazole in patients with pityriasis versicolor. Treatment response will be assessed clinically and mycologically to determine comparative outcomes.

DETAILED DESCRIPTION:
Pityriasis versicolor is a superficial fungal infection caused by Malassezia species and is commonly treated with topical antifungal agents. Ketoconazole is a conventional treatment, while luliconazole is a newer topical antifungal with potent activity against fungal organisms. This randomized controlled trial is designed to compare the clinical and mycological efficacy, safety, and tolerability of topical luliconazole versus topical ketoconazole in patients diagnosed with pityriasis versicolor. Eligible participants will be randomly allocated into two treatment groups and followed for treatment response and adverse effects. The findings of this study may help determine a more effective topical treatment option for pityriasis versicolor.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with pityriasis versicolor.

Exclusion Criteria:

* Immunocompromised patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Clinical and mycological cure rate in pityriasis versicolor. | 4 weeks
  Proportion of participants achieving both clinical and mycological cure.
Clinical and mycological cure | 4 weeks after completion of treatment
  Proportion of participants achieving both clinical and mycological cure

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared, as it is a small, single center based study. aggregate forms will be used to analyze the results. To ensure patients confidentiality data sharing is limited. Beyond the stated study object the dataset will not be used for any secondary purpose.

REFERENCES:
- See also: Related Info — https://ijhcr.com/index.php/ijhcr/article/download/4172/2894/6132